CLINICAL TRIAL: NCT05473910
Title: A Controlled Multi-Arm Phase 1 Umbrella Study Evaluating the Safety and Feasibility of T-Cell Receptor Engineered Donor T-Cells Targeting HA1 (TSC-100) or HA2 (TSC-101) in HLA-A0201 Positive Patients Undergoing Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: A Study of TSC-100 and TSC-101 in AML, ALL and MDS in Patients Undergoing Allogeneic Peripheral Blood Stem Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TScan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSCAN-001
Record Dates: First submitted 2022-07-11; First posted 2022-07-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: AML; Myelodysplastic Syndromes; ALL, Adult
Keywords: HA-1; HA-2; TSC-100; TSC-101; AML; MDS; ALL; Adoptive Cell Therapy; T-cell receptor; T lymphocyte; TCR-engineered T cells; bone marrow transplant; haploidentical; allogeneic stem cell transplant; BMT; Reduced Intensity Conditioning; RIC; HSCT; Hematopoietic stem cell transplantation; ALLOHA; Mismatched unrelated donors MMUD
MeSH Terms: conditions — Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TSC-100 Treatment Arm (Experimental): HA-1 positive patients
  Interventions: Drug: SOC + TSC-100
- TSC 101 Treatment Arm (Experimental): HA-1 negative and HA-2 positive patients
  Interventions: Drug: SOC + TSC-101
- Standard of Care or Control arm (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Drug: SOC + TSC-100 — HA-1 positive
  Arms: TSC-100 Treatment Arm
Drug: SOC + TSC-101 — HA-2 positive or HA-1 negative
  Arms: TSC 101 Treatment Arm
Other: Control — SOC alone
  Arms: Standard of Care or Control arm

SUMMARY:
This is a multi-center, non-randomized, concurrent controlled, multi-arm, Phase 1 interventional, open-label, biologic assignment-based umbrella study evaluating the feasibility, safety and preliminary efficacy of an escalating dose regimen of up to 2 doses of TSC-100 and TSC-101 in patients with AML, MDS, or ALL following HCT from a haploidentical donor, MMUD, or MUD

DETAILED DESCRIPTION:
A multi-center, non-randomized, controlled, multi-arm, Phase 1 interventional, open label, biologic assignment-based umbrella study is planned to evaluate the feasibility, safety, and preliminary efficacy of repeated dose regimen of TSC-100 and TSC-101 (TSC-100 and TSC-101 is a genetically engineered, donor-derived T cell targeting HA-1 and HA-2 respectively) in patients with AML, MDS, or ALL following HCT from a haploidentical donor, MUD, or MMUD.

The primary objective of this study is to investigate the safety of single and repeated dosing of TSC-100 and TSC-101 in HLA A*02:01 positive patients undergoing haploidentical allogeneic peripheral blood hematopoietic cell transplantation and determine the optimally tolerated dose range. The primary endpoints are: (1) incidence of dose-limiting toxicities (DLTs), and (2) incidence of adverse events (AEs) and serious AEs (SAEs) of TSC-100 and TSC-101 combined with the standard of care (SOC) compared with the SOC alone at 2 years of follow-up. The study will also investigate the efficacy of TSC-100 and TSC-101 combined with the SOC compared with that of the SOC alone to treat the study population and assess the immunogenicity of TSC-100 and TSC-101.

Depending on the HLA type and minor antigen positivity, patients will receive either TSC-100 or TSC-101 combined with the SOC or only SOC. TSC-100 or TSC-101 will be administered intravenously. Standard of care will include reduced intensity conditioning (RIC), hematopoietic cell infusion, and acute graft-versus-host disease (GvHD) prophylaxis. Patients will undergo one of the following RIC regimens, following standard institutional procedures: fludarabine+cyclophosphamide+total body irradiation, fludarabine+melphalan+/-total body irradiation, thiotepa+busulfan+fludarabine or flurdarabine+melphalan+thiotepa. In addition, patients may receive other supportive care measures and infectious prophylaxis as necessary, according to institutional guidelines or standards.

Successive cohorts of patients in the treatment arms will be started according to an interval 3+3 (i3+3) dose escalation design. Once the RP2D is identified, up to 20 additional patients may be enrolled at the RP2D. Dose escalations to the next cohort of TSC-100 and TSC-101 will be considered after the safety review committee (SRC) establishes reasonable safety for all patients enrolled into the current cohort. The safety and necessity of repeat dosing will also be determined by the SRC.

The safety data for all patients that received at least one dose of TSC-100 or TSC-101 in the treatment arms will be included in the safety assessment to proceed to the next dosing level and the dose escalation meeting will occur when the last patient in the cohort completes the 40-day DLT evaluation period. Depending on the number of DLTs observed, the range of patients that could be enrolled in the dose escalation stage of this i3+3 study is 35 to 300, including patients in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years at the time of signing the informed consent.
* Eastern Cooperative Oncology Group (ECOG)-PS ≤ 2 at the time of the screening visit.
* Contraceptive use by male and female participants must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male Participants:
* A male participant must agree to use a highly effective contraceptive as detailed in Appendix 4 of this protocol during the intervention period and for at least 12 months after the last dose of study intervention and refrain from donating sperm during this period.
* Female Participants:
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a woman of childbearing potential (WOCBP) OR
* A WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 12 months after the last dose of study intervention.
* Preparing to undergo allogeneic HCT for either of the following:
* AML
* MDS
* ALL
* Participants in the treatment arms must express HLA-A*0201. Participants in the control arm may express any HLA type.
* Having the HA1+/- or HA-1+/+ (HA-1 positive) genotype to be eligible for TSC-100 treatment.
* Having the HA2+/- HA-2+/+ (HA-2 positive) genotype to be eligible for TSC-101 treatment.
* Having a haploidentical donor, MMUD, or MUD for HCT who is adequately HLA-matched by institutional standards and meets the donor inclusion criteria.
* Considered to be clinically indicated for haploidentical donor, MMUD, or MUD transplantation at the discretion of the treating investigator.
* Considered to be clinically indicated for RIC at the discretion of the treating investigator.
* Considered to be clinically indicated for peripheral blood stem cell transplantation at the discretion of the treating investigator.
* Organ function parameters for transplant eligibility are met per institutional standards.
* Capable of giving signed informed consent - which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Participants must provide consent for mandatory study procedures including bone marrow biopsy and blood sampling for research analyses in the ICF.
* Participants must agree to participate in long-term follow-up for up to 15 years post initial product treatment if they are enrolled in the study and receive the investigational Tcell infusion.

Donor Inclusion Criteria :

* Male or female aged ≥ 18 years at the time of signing the informed consent.
* Able to undergo peripheral blood stem cell (PBSC) collection and up to 2 rounds of leukapheresis (for TSC-100 or TSC101 manufacturing for treatment arms only, and f for stem cell collection for both treatment arms and the control arm).
* Donors matched to TSC-100 participants should be HA-1-/- (negative) and/or negative for all HLA-A*02 alleles
* Donors matched to TSC-101 participants should be negative for all HLA-A*02 alleles
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Medical or psychological conditions that would make the participant an unsuitable candidate for cell therapy including another concurrent uncontrolled malignancy or active CNS disease.
* The presence of organ toxicities will not necessarily exclude participants from enrolling on the protocol at the discretion of the PI; however, a delay in the infusion of HA1/HA2 TCRT cells may be required at the discretion of the treating investigator
* Participants with levels of donor-specific HLA antibodies that are considered by the treating investigator to be high enough to warrant desensitization protocols and who have no alternate donors.
* Participants who meet inclusion criteria for TSC-101 but who are also positive for HLAA*02:07.
* Participants with evidence of clinically significant infection or uncontrolled viral r reactivation of cytomegalovirus (CMV), Epstein-Barr virus (EBV), Adenovirus, BK virus (BKV), or human herpesvirus 6 (HHV-6).
* Participants with active cardiac disease, defined as:
* Uncontrolled or symptomatic angina within the past 3 months.
* History of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, torsades de pointes). Atrial fibrillation with controlled ventricular response on treatment is not an exclusion.
* Myocardial infarction < 3 months from study entry.
* Uncontrolled or symptomatic congestive heart failure.
* Prior allogeneic HCT.
* Participants who have a history of hypersensitivity to murine proteins.
* Enrollment on a concomitant trial with a novel investigational agent.
* Use of anti-thymocyte globulin, alemtuzumab, or other in vivo T-cell depleting agents from Day -14 through end of study.

Donor Exclusion Criteria :

* Donors for TSC-100 positive for any HLA-A*02 allele would be excluded unless they are HA-1 negative. If donors with any HLA-A*02 allele are considered for patients eligible for TSC-100, the donor would undergo HA-1 testing to ensure that the donor is HA-1 negative (40% probability).
* Donors for TSC-101 positive for any HLA-A*02 allele are excluded regardless of HA- 2 status.
* Donors who test positive for any of the following: HIV-1, HIV-2, human T-lymphotropic virus (HTLV)-1, HTLV-2 seropositive or with active hepatitis B or hepatitis C virus infection, syphilis, West Nile virus through central lab testing. Donors who screen positive for risk of CreutzfeldtJakob disease or Zika virus infection using donor history questionnaires will also be excluded. Donors with evidence of past CMV or EBV infections will be allowed.
* Related donor residing outside of the United States of America (USA). If the donor screening, testing and leukapheresis can be performed at the same site where the participant is being treated, the donor is considered eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities | two years
  Number of DLTs observed in patients compared to the control arm
Occurrence of adverse events | two years
  Number of adverse events in patients compared to control arm

SECONDARY OUTCOMES:
Comparison of disease free survival in patients versus the control arm | 6 months
  Disease-free survival in patients versus the control arm at 6 months, defined as the time from date of transplant to death or relapse/progression, whichever comes first. Participants alive and disease free will be censored at the last follow-up.
Comparison of disease free survival in patients versus the control arm | 12 months
  Disease-free survival in patients versus the control arm at 12 months, defined as the time from date of transplant to death or relapse/progression, whichever comes first. Participants alive and disease free will be censored at the last follow-up.
Disease-free survival in patients versus the control arm at 18 months, defined as the time from date of transplant to death or relapse/progression, whichever comes first. Participants alive and disease free will be censored at the last follow-up. | 18 months
  Disease-free survival at Month 18 defined as the time from date of transplant to death or relapse/progression, whichever comes first. Participants alive and disease free will be censored at the last follow-up.
Comparison of disease free survival in patients versus the control arm | 24 months
  Disease-free survival in patients versus the control arm at 24 months, defined as the time from date of transplant to death or relapse/progression, whichever comes first. Participants alive and disease free will be censored at the last follow-up.
Comparison of relapse rates between patients and control arm | 6 months
  Relapse rates in patients versus the control arm at 6 months. Relapse is defined by either morphological or cytogenetic evidence of acute leukemia or MDS consistent with pre-transplant features, or radiologic evidence of lymphoproliferative disorders, documented or not by biopsy.
Comparison of relapse rates between patients and control arm | 12 months
  Relapse rates in patients versus the control arm at 12 months. Relapse is defined by either morphological or cytogenetic evidence of acute leukemia or MDS consistent with pre-transplant features, or radiologic evidence of lymphoproliferative disorders, documented or not by biopsy.
Comparison of overall survival between patients and control arm | Up to 2 years
  Overall survival between patients versus the control arm, defined as the time interval between the date of transplant and death from any cause. Surviving participants will be censored at the last follow up.
Anti TSC-100 antibodies | 2 years
  Presence and concentration of anti TSC-100 antibodies.
Anti TSC-101 antibodies | 2 years
  Presence and concentration of anti TSC-101 antibodies.

OTHER OUTCOMES:
Analysis of donor chimerism | 60 days
  Analysis of donor hematopoietic chimerism evaluated in bone marrow, whole unfractionated blood, or blood cell fractions, including CD3 and CD33 subsets.
Analysis of donor chimerism | 100 days
  Analysis of donor hematopoietic chimerism evaluated in bone marrow, whole unfractionated blood, or blood cell fractions, including CD3 and CD33 subsets.
Analysis of MRD | 60 days
  MRD status in bone marrow biopsies at Day 60
Analysis of MRD | 100 days
  MRD status in bone marrow biopsies at Day 100
Analysis of MRD | 180 days
  MRD status in bone marrow biopsies at Day 180.
HA-1 persistence | 2 years
  Persistence of HA1 TCRT cells in the peripheral blood and bone marrow, measured in bone marrow or whole unfractionated blood by a central laboratory flow cytometric assay.
HA-2 persistence | 2 years
  Persistence of HA2 TCRT cells in the peripheral blood and bone marrow, measured in bone marrow or whole unfractionated blood by a central laboratory flow cytometric assay.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Matzko, MD, Study Director — Tscan Therapeutics
Locations (15):
- United States (15):
  - City of Hope, Duarte, California
  - Yale, New Haven, Connecticut
  - Memorial Healthcare System, Hollywood, Florida
  - Northside Hospital, Atlanta, Georgia
  - John Hopkins University, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - Mount Sinai, New York, New York
  - University North Carolina, Chapel Hill, North Carolina
  - UPenn, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Froedert and Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No